CLINICAL TRIAL: NCT00865254
Title: Prize Reinforcement for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, David Ledgerwood, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDA021839A; R21DA021839 (NIH); 1R21DA021839-01 (NIH)
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Nicotine Dependence
Keywords: Nicotine Dependence; Smoking; Smoking Cessation; Contingency Management
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Traditional Contingency Management (Experimental): Standard treatment plus prize based contingency management.
  Interventions: Behavioral: Traditional Contingency Management
- Early Enhanced Contingency Management (Experimental): Prize based contingency management with enhanced magnitude early in treatment and reduced magnitude later in treatment.
  Interventions: Behavioral: Early Enhanced Contingency Management
- Standard Treatment (Active Comparator): Counseling and monitoring of smoking cessation.
  Interventions: Behavioral: Standard Treatment

INTERVENTIONS:
Behavioral: Standard Treatment — Brief counseling for smoking cessation followed by continued brief supportive sessions and frequent monitoring of smoking cessation efforts.
  Arms: Standard Treatment
Behavioral: Traditional Contingency Management — Prize based contingency management condition in which participants have the chance to win incentives (prizes) when they provide biological test results (expired carbon monoxide and cotinine) that are negative for recent smoking. Prize draws result in incentives on an intermittent schedule (50% of draws are prizes). Participants are also provided with brief counseling for smoking cessation followed by continued brief supportive sessions and frequent monitoring of smoking cessation efforts.
  Arms: Traditional Contingency Management
Behavioral: Early Enhanced Contingency Management — Prize based contingency management condition in which participants have the chance to win incentives (prizes) when they provide biological test results (expired carbon monoxide and cotinine) that are negative for recent smoking. Prize draws result in incentives on an intermittent schedule (100% of draws are prizes in week 1; 33% are prizes in weeks 2-4). Participants are also provided with brief counseling for smoking cessation followed by continued brief supportive sessions and frequent monitoring of smoking cessation efforts.
  Arms: Early Enhanced Contingency Management

SUMMARY:
Nicotine dependence is prevalent in society, cigarette smoking is associated with several known health risks, and most dependent individuals find it very difficult to stop smoking cigarettes. The present study will test the efficacy of a behavioral smoking cessation treatment, prize-based contingency management, that has not undergone rigorous study with respect to smoking, it but has demonstrated efficacy in reducing use of other substances (e.g. cocaine). If efficacious, prize-based contingency management would add to our repertoire of efficacious smoking cessation treatments.

DETAILED DESCRIPTION:
Contingency management (CM) treatments are efficacious in reducing substance use. A relatively new approach, called prize-based CM, which uses prizes to reinforce substance abstinence, is effective in decreasing certain types of substance use, but its efficacy has not been evaluated in the treatment of cigarette smoking. One purpose of the current study is to assess the efficacy of a prize reinforcement intervention for reducing cigarette smoking. A second purpose is to test the differential efficacy of two schedules of reinforcement, using cigarette smoking as an exemplar. We will randomly assign 110 patients to one of three conditions: 1) Standard treatment; 2) Traditional prize reinforcement; or 3) Early-treatment enhanced prize reinforcement. Patients in each condition will receive counseling for their smoking based on current standard of care guidelines. All patients will participate in a one-week baseline period, followed by a four-week intervention. Throughout both phases, each patient will meet with a research assistant twice daily to provide carbon monoxide (CO) samples. Patients in the prize reinforcement conditions will earn the chance to win prizes when they provide negative CO samples (i.e., < 6ppm). They will also earn bonus draws if they provide negative cotinine samples (i.e., <100ng/ml) after weekends. Patients in the Traditional CM condition will have at least a 50% chance of winning a prize for each negative sample with escalating chances for successive negative samples. Patients in the Enhanced condition will have the opportunity to earn the same overall number of draws and magnitude of reinforcement, but the schedule of reinforcement will differ. For the first week of the CM phase, these patients will have a 100% chance of winning prizes, but in the latter 3 weeks, overall probability of reinforcement will be decreased to 34%. Patients will also undergo 2- and 6-month follow-up assessments. Primary outcome measures will be longest duration of continuous abstinence and mean number of days of abstinence. We predict that the prize reinforcement will reduce cigarette smoking to a greater extent than standard treatment. We also predict that the Enhanced CM condition will lead to greater reductions in cigarette smoking relative to the Traditional CM condition, and that these changes may result in longer sustained abstinence from smoking throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. A current Fagerstrom scale score of 6 or greater;
2. Age 13 years old or older (Under age 18, parental consent is required);
3. Able to read and understand English.

Exclusion Criteria:

1. Have current severe, uncontrolled psychiatric disorders (i.e., acute suicidality or psychosis);
2. Have current substance dependence, other than nicotine or caffeine dependence;
3. Are in recovery for pathological gambling; or
4. Are already participating in other behavioral or medication smoking cessation programs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Expired Carbon Monoxide | Baseline and treatment phases, 2-mont and 6-month follow up.

SECONDARY OUTCOMES:
Self-reported smoking. | Baseline, throughout treatment, 2-month and 6-month follow up.
Cotinine levels. | Baseline, throughout treatment, 2-month and 6-month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: David M Ledgerwood, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Jefferson Avenue Research Clinic, Detroit, Michigan, United States

REFERENCES:
- [Derived] Reid HH, Ledgerwood DM. Depressive symptoms affect changes in nicotine withdrawal and smoking urges throughout smoking cessation treatment: Preliminary results. Addict Res Theory. 2016;24(1):48-53. doi: 10.3109/16066359.2015.1060967. Epub 2015 Jun 26. PMID 27547173